CLINICAL TRIAL: NCT06135948
Title: Impact of Increasing Levothyroxine Dose in Ramadan for UAE Patients With Hypothyroidism: a Randomized Controlled Trial
Brief Title: Impact of Increasing Levothyroxine Dose in Ramadan for UAE Patients With Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emirates Health Services (EHS) (Other Government)
Collaborators: University of Sharjah (Other)
Responsible Party: Principal Investigator, Dr. Nawal Almutawa,MD,FCCE,FACE,EMPA, Principle investigator,Dr. Nawal Al mutawa, Consultant I.M, Endocrinologist & Dialectologist, Head of Department of Endocrinology & Dialectology, Emirates Health Service, UAE MD, I.M board BIM (FCCE (FACE), (EMPA) Past Medical Director, Emirates Health Services (EHS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXL-THYROXINE2023
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: L-thyroxine

STUDY DESIGN:
Intervention Model Description: The present study is an open-label, two-arm parallel groups, randomized controlled clinical trial that included Emirati patients with hypothyroidism who attended the Family Promotion Centre, Endocrinology Clinic, regularly. Eligible participants (n = 103) were randomly allocated to the treatment group (patients who received an increased dose of L-thyroxine, 25 mcg, n = 50) and the control group (patients who received standard/regular dose of L-thyroxine, n = 46). Both groups attended 5 visits before, during, and after Ramadan. Several tests were conducted including thyroid function, lipid profile, HbA1c, and Vitamin D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Hypothyroidism patients who received an increased dose of L-thyroxine, 25 mcg, n = 50
  Interventions: Drug: Extra dose of L-thyroxine, 25 mcg during Ramadan
- Control Group (No Intervention): Hypothyroidism patients who received standard/regular dose of L-thyroxine, n = 46

INTERVENTIONS:
Drug: Extra dose of L-thyroxine, 25 mcg during Ramadan — Extra dose of L-thyroxine, 25 mcg during the month of Ramadan
  Arms: Intervention Group

SUMMARY:
The study aims to compare the mean change in Thyroid Stimulating Hormone (TSH) levels among patients with hypothyroidism treated with an increased dose of L-thyroxine (treatment group) versus standard/regular dose of L-thyroxine (control group) during the month of Ramadan.

DETAILED DESCRIPTION:
The present study is an open-label, two-arm parallel groups, randomized controlled clinical trial that included Emirati patients with hypothyroidism who attended the Family Promotion Centre, Endocrinology Clinic, regularly. Eligible participants (n = 103) were randomly allocated to the treatment group (patients who received an increased dose of L-thyroxine, 25 mcg, n = 50) and the control group (patients who received standard/regular dose of L-thyroxine, n = 46). Both groups attended 5 visits before, during, and after Ramadan. Several tests were conducted including thyroid function, lipid profile, HbA1c, and Vitamin D.

ELIGIBILITY:
The inclusion criteria for participants will include:

1. Male and female patients with primary hypothyroidism.
2. Patients with stable TSH
3. Aged between 18 and 70 years.
4. Patients regularly fasting for at least 25- 30 days during Ramadan.
5. Emirati nationals (100% health care coverage)

Exclusion Criteria:

1. Patients with any end organ damage
2. Pregnant or Breast-feeding women
3. Thyroid cancer
4. Patients not adhering to initial thyroxine medications.
5. Those receiving proton pump inhibitory therapy, dietary fiber, bile acid sequestrates, ferrous sulfate, sucralfate, calcium carbonate, aluminum-containing antacids, phosphate binders, and raloxifene.
6. Disease interferes with thyroxine absorption, coeliac disease, inflammatory bowel disease, lactose intolerance as well as Helicobacter pylori (H. pylori) infection and atrophic gastritis,
7. Several other factors cause treatment failures such as fiber-rich food, soy protein, grapefruit, and aluminum antacids, which interfere with Thyroxine absorption. In addition to calcium carbonate and ferrous sulfate.
8. Patients were diagnosed with cardiovascular disorders, including angina, coronary artery disease, and hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Effects of an extra dose of L-thyroxine during the month of Ramadan | 3 months
  to compare the mean change in Thyroid Stimulating Hormone (TSH) levels among patients with hypothyroidism treated with an increased dose of L-thyroxine (treatment group) versus standard/regular dose of L-thyroxine (control group) during the month of Ramadan.

CONTACTS AND LOCATIONS:
Locations (1):
- Family Promotion Centre, Endocrinology Clinic, Sharjah city, United Arab Emirates